CLINICAL TRIAL: NCT05233930
Title: Does an Augmented Reality-based Navigation System in Total Knee Arthroplasty Allow a Better Alignment of the Lower Limb and Does it Improve Functional Results ? An Equivalence, Monocentric, Prospective and Randomized Study
Brief Title: Total Knee Arthroplasty and Augmented Reality-based Navigation System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TKA and augmented reality; 2021-A02549-32 (Other: ANSM)
Record Dates: First submitted 2022-01-18; First posted 2022-02-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Gonarthrosis
Keywords: TKR: total knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — tokaratoxin 2

STUDY DESIGN:
Intervention Model Description: Randomised, double-arms, parallel, open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TKR with augmented reality-based navigation system. (Experimental): This technology offers the orthopedic surgeon intraoperative assistance in positioning the implants with the help of a pair of augmented reality glasses. The cutting planes are oriented with respect to the mechanical axes calculated according to anatomical landmarks acquired with a pointer. The connected glasses calculate precisely the 3D coordinates of the instruments thanks to the analysis of their specific markers (QR-Code), filmed by the integrated camera. The navigation information is displayed in the surgeon's field of vision, who interacts with the application thanks to the glasses' accelerometers.
  Interventions: Procedure: TKR with augmented reality-based navigation system
- TKR with traditional mechanically aligned technique. (Active Comparator): TKR with traditional mechanically aligned technique will be performed according to local practice and standard guidelines.
  Interventions: Procedure: TKR with traditional mechanically aligned technique

INTERVENTIONS:
Procedure: TKR with augmented reality-based navigation system — Surgery
  Arms: TKR with augmented reality-based navigation system.
Procedure: TKR with traditional mechanically aligned technique — As per local practice and standard guidelines.
  Arms: TKR with traditional mechanically aligned technique.

SUMMARY:
The purpose of Total Knee Replacement (TKR) is to remove worn cartilage surfaces and replace them with artificial parts of the same shape. TKR can be used in cases of osteoarthritis, inflammatory rheumatism, bone necrosis of the knee or following malformative or traumatic sequelae.

Implant alignment is paramount in TKR and the last years have seen a proliferation of alignment techniques following the introduction of computer and robotic-assisted surgery. Among Computer-assisted surgery, the augmented reality-based navigation system can be an option to improve accuracy in orthopaedic surgery.

The hypothesis of this study is: the use of augmented reality-based navigation system allows a prosthesis alignment and positioning that is at least as good as with the traditional mechanically aligned technique, and therefore improves knee functional results. This study also aims at assessing the cost-effectiveness of this new technology.

DETAILED DESCRIPTION:
In this randomised study, TKR will be performed either with the traditional mechanically aligned technique or with an augmented reality-based navigation system using Knee+ technology.

Knee+ is a Class Im software medical device (European classification, Directive 93/42/EEC, Annex IX) and obtained CE Mark 0459 in May 2020.

This technology is used in total knee replacement procedures, and offers the orthopedic surgeon intraoperative assistance in positioning the implants with the help of a pair of augmented reality glasses. The cutting planes are oriented with respect to the mechanical axes calculated according to anatomical landmarks acquired with a pointer. The connected glasses calculate precisely the 3D coordinates of the instruments thanks to the analysis of their specific markers (QR-Code), filmed by the integrated camera. The navigation information is displayed in the surgeon's field of vision, who interacts with the application thanks to the glasses' accelerometers.

ELIGIBILITY:
Inclusion Criteria:

1. Gonarthrosis on a varum knee requiring a Total Knee Replacement
2. Female or male, 18 years of age or older
3. Affiliation to a social security scheme
4. Patient has been informed of the study and has signed an informed consent form

Exclusion Criteria:

1. Osteonecrosis,
2. Post traumatic osteoarthritis with femoral or tibial callus,
3. History of tibial or femoral osteotomy,
4. Valgum knee,
5. Isolated patellofemoral osteoarthritis,
6. Significant hip dysplasia or other excessive pelvic deformity,
7. Patient already equipped with medical devices that may conflict with the instrumentation required for augmented reality navigation,
8. Pregnant or breastfeeding women,
9. Patients under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Radiographic evaluation of the Hip-Knee-Ankle (HKA) angle | 2 months after surgery
  the Hip-Knee-Ankle (HKA) angle is measured on weight bearing pangonogram.

SECONDARY OUTCOMES:
Evaluation of long-term lower limb alignment between the two procedures | 1 year after surgery
  Radiographic evaluation of the Hip-Knee-Ankle (HKA) angle on lower limb pangonogram at 1 year after surgery
Evaluation of the success of the procedure | 2 months after surgery
  The success of the procedure is defined by an HKA angle of 180°
Assessment of lower limb alignment variability between the two procedures. | 2 months and1 year after surgery
  Radiographic evaluation of the Hip-Knee-Ankle (HKA) angle on lower limb pangonogram at 2 months and 1 year after surgery.
Evaluation of radiological measurements between the two procedures | 2 months and1 year after surgery
  Evolution of the following radiological parameters at 2 months and 1 year post-surgery:
  Femoral valgus Tibial varus Posterior tibial slope Flessum of the femoral implant Patellar tilt
Evaluation of the knee score between the two procedures | 2 months and1 year after surgery
  Evolution of the knee score at 2 months and 1 year postoperatively measured by the Knee Society Score (KSS). The KSS is a widely used clinician-assessed outcome score with good published validity data. The clinical part (Knee Score) of the KSS covers pain, range of motion, alignment and stability. The Function Score of the KSS covers patient mobility (walking distance and stairs) and potential walking aids. The KSS scoring scale ranges from 0 to 100 points for each part, with higher scores indicating less severe impairment.
Quality of life assessment between the two procedures | 2 months and1 year after surgery
  Change in quality of life at 2 months and 1 year measured by the Short Form-12 (SF-12) questionnaire.
  The SF-12 is a standardized self-questionnaire for measuring quality of life.The SF-12 is the shortened version of the SF-36.
  The SF-12 is made up of eight subscores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a scale from 0 to 100 on the assumption that each question has the same weight. The lower the score, the greater the handicap. The higher the score, the lower the handicap, i.e. a score of zero equals maximum handicap and a score of 100 equals zero handicap.
Evaluation of knee pain between the two procedures | From day 0 to day 5 ; Once a week during 1 month ; at 2 months ; at 3 months and 1 year after surgery
  Evolution of pain every day between D0 (postoperative) and D5, then once a week during the first month, then at 2 months, 3 months and at 1 year postoperative measured by a visual analog scale (VAS).
  The visual analog scale (VAS) for pain is a pain self-assessment tool. The patient defines his pain on a line 10cm long. The distance (in millimeters) from the left extremity defines the pain. The value zero corresponds to the lower limit defining the absence of pain and 100 to the upper limit corresponding to "the worst pain imaginable".
Evaluation of the hemoglobin level between the two procedures | From day 1 to day 3 after surgery
  Evolution of the hemoglobin level at D1 and D3
Evaluation of the Average Length of Stay between the two procedures | From the day of surgery at the time of hospital discharge up to 1 day
  The Average Length of Stay will be evaluated in days from the hospital's entry and exit records.
Evaluation of the postoperative complications rate between the two procedures | During 1 year post-operative
  Occurrence of a thromboembolic complication (yes/no) during the 1-year post-operative follow-up.
  Occurrence of a surgical site infection (yes/no) during the 1-year post-operative follow-up.
  Occurrence of wound healing problems (yes/no) during the 1-year post-operative follow-up
Evaluation of the Quality-Adjusted Life Years (QALY) between the two procedures | At 1 year
  EQ-5D questionnaire at 1 year and collection of all costs during the first postoperative year.

OTHER OUTCOMES:
Radiographic assessment | At 2 months after surgery
  The primary endpoint of this research will be radiographic assessment of the Hip-Knee-Ankle (HKA) angle on weight-bearing lower extremity pangonometry at 2 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Dalat, MD, Principal Investigator — Centre Médico-Chirurgical de Tronquières
Locations (1):
- Centre Médico-Chirurgical de Tronquières, Aurillac, France

REFERENCES:
- [Background] Panjwani TR, Mullaji A, Doshi K, Thakur H. Comparison of Functional Outcomes of Computer-Assisted vs Conventional Total Knee Arthroplasty: A Systematic Review and Meta-Analysis of High-Quality, Prospective Studies. J Arthroplasty. 2019 Mar;34(3):586-593. doi: 10.1016/j.arth.2018.11.028. Epub 2018 Dec 2. PMID 30611520
- [Background] Cheng T, Pan XY, Mao X, Zhang GY, Zhang XL. Little clinical advantage of computer-assisted navigation over conventional instrumentation in primary total knee arthroplasty at early follow-up. Knee. 2012 Aug;19(4):237-45. doi: 10.1016/j.knee.2011.10.001. Epub 2011 Nov 29. PMID 22130355
- See also: Computer-assisted navigation system (CAS) in total knee arthroplasty (TKA) has been shown to improve mechanical alignment and prosthesis positioning as compared to conventional TKA. — https://pubmed.ncbi.nlm.nih.gov/30611520/
- See also: Even though computer-assisted navigation systems have been shown to improve the accuracy of implantation of components into the femur and tibia, long-term results are lacking — https://pubmed.ncbi.nlm.nih.gov/22130355/